CLINICAL TRIAL: NCT04579419
Title: Injection Site Pain, Onset and Duration of Action of Botulinum Toxin Reconstituted in Normal Saline With and Without Sodium Bicarbonate; A Prospective, Single Center, Randomized, Double-Blind Interventional Study
Brief Title: Injection Site Pain Botulinum Toxin Reconstituted in NS With and Without Sodium Bicarbonate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, Leen Hijazi, Medical Intern, King Abdulaziz Medical City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC19/371
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Wrinkle
MeSH Terms: interventions — Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate (Experimental)
  Interventions: Drug: Sodium Bicarbonate
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Sodium Bicarbonate — Botulinum Toxin diluted in Sodium Bicarbonate
  Arms: Sodium Bicarbonate
Drug: Normal Saline — 0.9 NaCl
  Arms: Normal Saline

SUMMARY:
This study was designed to investigate the effects of botulinum toxin type A injections diluted with the mixture of sodium bicarbonate (SB) and normal saline (NS) on pain reduction, onset of action and duration of action.

This is a prospective, randomized, double-blind clinical study, which included 30 female patients (age>25). The patients were randomized to receive botulinum toxin (BT) injections diluted with NS and SB on one side of the face and saline control injections on the other side. Pain severity was assessed using visual analogue scale. The onset and duration of action were recorded according to the patients' subjective opinions after 1 week and 3 months, respectively. The study was approved with an IRB (Institutional Review Board) number of RC19/371.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient who is in good health and has moderate dynamic forehead and glabellar wrinkles.

Exclusion Criteria:

* • Patients <25 years old

  * Presence of neuromuscular disease or intake of drugs affecting muscle tone.
  * Any active infection in the treatment area.
  * Patients receiving anticoagulation or had a diagnosis of bleeding disorders.
  * Any patient who had undergone the following treatments to the forehead area in the past 6 months: botulinum toxin injections, ablative laser procedures, radiofrequency device treatments, ultrasound device treatments, or medium to deep chemical peels.
  * Any patient who had temporary soft-tissue augmentation material to the forehead area in the past 12 months, semi permanent soft-tissue augmentation material in the past 2 years, or permanent soft-tissue augmentation material at any point in the past.
  * Any patient with prior facial cosmetic surgical procedures such as eyebrow-lifts, blepharoplasties, and rhytidectomies.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-09 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2020-08-09 (Actual)

PRIMARY OUTCOMES:
Injection site pain | Immediately after the injections
  Pain severity was assessed using Visual Analogue Scale (VAS).The VAS score ranged from 0 to 10, with 0 representing no pain and 10 the greatest imaginable pain. Higher scores indicated worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Saudi Arabia